CLINICAL TRIAL: NCT07079111
Title: 3D Printed Occlusal Splints for Intraoperative Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00515012
Record Dates: First submitted 2025-07-21; First posted 2025-07-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Malocclusion, Angle Class I; Malocclusion, Angle Class II; Malocclusion, Angle Class III
Keywords: malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class I; Malocclusion, Angle Class II; Malocclusion, Angle Class III; Malocclusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Industry made splint (Experimental): Occlusal splints will be 3D printed by industrial third party
  Interventions: Device: Industry made occlusal splint
- In House made splint (Experimental): In house 3D printed occlusal splint
  Interventions: Device: Formlabs 3D printed occlusal splint

INTERVENTIONS:
Device: Formlabs 3D printed occlusal splint — In house 3D printed occlusal splint with Formlabs printer
  Arms: In House made splint
Device: Industry made occlusal splint — Industry made occlusal splint
  Arms: Industry made splint

SUMMARY:
A 3D printed intraoperative occlusal splint is a custom-made biocompatible resin guide that allows surgeons properly align a patient's upper and lower dentition during surgery. This alignment further places maxilla and mandible into proper position. An occlusal splint contains outlines maxillary and mandibular dentition allowing the teeth to lock into place with correct alignment.

At Johns Hopkins, traditionally hand-made and industry-made 3D printed splints have been used safely. However, prior studies have demonstrated the ability of in-house 3D prints to save time and money compared to industry. In-house models are similarly produced with FDA-clear, biocompatible resin for 3D printing, and maintain equivalent safety for patients compared to industry-made models.

DETAILED DESCRIPTION:
Treatment of dentofacial deformities requires restoration of occlusion. Occlusal splints stabilize the jaws intraoperatively to restore occlusion, which improve functions such as mastication, speech, breathing, and appearance.

Orthodontic resins and denture material have been used to fabricate dental splints due to the biocompatibility nature and ease of use. These materials, throughout the years, have been found to have structural stability, used for various purposes including nightguards, occlusal splints, etc. In recent years with the advanced of computer automated design (CAD/CAM), these splints have been outsourced to industry manufacturers.

Industry-made printed splints are costly and time-consuming, highlighting the need for faster, more affordable solutions. In-house printed splints have demonstrated consistent uniformity with negligible differences in shape to the source files. The investigators hypothesize that in-house printed models will be at least as effective as industry-made models in the application of acute craniofacial trauma while decreasing costs and production time.

This study evaluates the feasibility and benefits of in-house 3D printed occlusal splints. By using the same printers and biocompatible resin as industry manufacturers12, in-house splints maintain patient safety, while reducing hospital stay durations, lowering infection rates, and increasing hospital turnover. This approach could improve surgical efficiency and patient outcomes, offering a cost-effective alternative in mandibular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age who require any orthognathic surgery (including, but not limited to, facial fracture reduction and fixation, mandibular or maxillary reconstruction, cranial vault reconstruction, mandibular osteotomies, maxilla osteotomies) at Johns Hopkins Hospital.

Exclusion Criteria:

* Patients who are non-English speaking.
* Surgeons who do not perform orthognathic surgery with occlusal splints.

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2030-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Time (hours) of delivery of models | Up to 1 year
  Time of delivery of in-house and industry made splint models.
Cost of production for oral splint models | Up to 1 year
  Cost of production of in-house and industry-made models
Surgeon satisfaction assessed by survey | Post surgery up to 1 month
  Surgeon satisfaction between industry-made and in-house 3D printed occlusal splints. Score range between 5-20. Higher score more satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Yang, MD, DDS, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: Yes
Once the project has been published, a workflow will be published alongside it.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Wezgowiec J, Malysa A, Szlasa W, Kulbacka J, Chwilkowska A, Zietek M, Wieckiewicz M. Biocompatibility of 3D-printed vs. thermoformed and heat-cured intraoral appliances. Front Bioeng Biotechnol. 2024 Oct 29;12:1453888. doi: 10.3389/fbioe.2024.1453888. eCollection 2024. PMID 39534672
- [Background] Beidas T, Light L, Carrico C, Kondor S, Ravi P, Rabinowitz YA. Printing outsourced orthognathic surgical splints in-house: a dimensional verification process for point-of-care printing. 3D Print Med. 2025 Jun 6;11(1):24. doi: 10.1186/s41205-025-00276-9. PMID 40478376
- [Background] Chen K, Kreh CC, Lin AY. In-House 3D Printing for Craniofacial Trauma: 7-Year Review. Ann Plast Surg. 2025 May 1;94(5S Suppl 3):S435-S440. doi: 10.1097/SAP.0000000000004281. PMID 40310006
- [Background] Shilo D, Capucha T, Krasovsky A, Blanc O, Emodi O, Haze A, Rachmiel A. Real-time Reconstruction of Comminuted Mandibular Fractures Using 3D Printing. Plast Reconstr Surg Glob Open. 2024 Mar 20;12(3):e5645. doi: 10.1097/GOX.0000000000005645. eCollection 2024 Mar. PMID 38510331
- [Background] DeBusk WT, Bhethanabotla RM, David AP, Heaton CM, Park AM, Seth R, Knott PD. Cost Comparison of Industry Versus In-House Three-Dimensional Printed Models for Microvascular Mandible Reconstruction. Facial Plast Surg Aesthet Med. 2025 Mar-Apr;27(2):157-162. doi: 10.1089/fpsam.2024.0172. Epub 2024 Nov 22. PMID 39574355
- [Background] Marschall JS, Oppenheim MA, Kushner GM. Can a Point-of-Care 3D Printing Workflow Produce Accurate and Successful Results for Craniomaxillofacial Trauma? J Oral Maxillofac Surg. 2024 Feb;82(2):207-217. doi: 10.1016/j.joms.2023.11.006. Epub 2023 Nov 10. PMID 38012957
- [Background] Ureel M, Bodere PJ, Denoiseux B, Corthouts P, Coopman R. Mandibular Reconstruction with Osseous Free Flap and Immediate Prosthetic Rehabilitation (Jaw-in-a-Day): In-House Manufactured Innovative Modular Stackable Guide System. Bioengineering (Basel). 2024 Dec 11;11(12):1254. doi: 10.3390/bioengineering11121254. PMID 39768072
- [Background] Kim E, Vishwanath N, Foppiani J, Escobar-Domingo MJ, Lee D, Francalancia S, Lin GJ, Woo AS, Lin SJ. Barriers of Three-Dimensional Printing in Craniofacial Plastic Surgery Practice: A Pilot Study and Literature Review. J Craniofac Surg. 2024 Jun 1;35(4):1105-1109. doi: 10.1097/SCS.0000000000010271. Epub 2024 May 10. PMID 38727233
- [Background] Oley MH, Oley MC, Sukarno V, Faruk M. Advances in Three-Dimensional Printing for Craniomaxillofacial Trauma Reconstruction: A Systematic Review. J Craniofac Surg. 2024 Oct 1;35(7):1926-1933. doi: 10.1097/SCS.0000000000010451. Epub 2024 Jul 3. PMID 38958985
- [Background] Gomez VJ, Martin-Gonzalez A, Zafra-Vallejo V, Zubillaga-Rodriguez I, Fernandez-Garcia A, Sanchez-Aniceto G. In-House Virtual Surgery Planning and 3D Printing for Head and Neck Surgery With Free Software: Our Workflow. Craniomaxillofac Trauma Reconstr. 2024 Dec;17(4):331-339. doi: 10.1177/19433875231211759. Epub 2023 Nov 15. PMID 39634570
- [Background] Gomez VJ, Martin-Gonzalez A, Zafra-Vallejo V, Zubillaga-Rodriguez I, Fernandez-Garcia A, Sanchez-Aniceto G. Controversies in point-of-care 3D printing for oncological and reconstructive surgery with free software in oral and maxillofacial surgery: European regulations, costs, and timeframe. Int J Oral Maxillofac Surg. 2024 Aug;53(8):650-660. doi: 10.1016/j.ijom.2024.01.005. Epub 2024 Jan 29. PMID 38290865
- [Background] ElShebiny T, Simon Y, Demko CA, Palomo JM. The uses of 3-dimensional printing technology in orthodontic offices in North America. Am J Orthod Dentofacial Orthop. 2024 Jul;166(1):76-80. doi: 10.1016/j.ajodo.2024.03.014. Epub 2024 Apr 26. PMID 38678454